CLINICAL TRIAL: NCT05351710
Title: A Randomized Controlled Trial of an Exposure-Based Treatment for Perfectionism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Professor of Psychology, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003084
Record Dates: First submitted 2022-04-24; First posted 2022-04-28 (Actual); Results first posted 2024-07-15 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Perfectionism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure-Based Treatment for Perfectionism (Experimental): This arm consists of a 2-week computerized, exposure-based intervention. Treatment sessions are completed every 2 days at home (8 treatment sessions total).
  Interventions: Behavioral: Exposure-Based Treatment for Perfectionism
- Stress Management Condition (Active Comparator): This arm consists of a 2-week, computerized, stress-management condition in which participants watch videos of health habits (e.g., nutrition, exercise, sleep) and relaxation videos. These sessions are completed every 2 days at home (8 sessions total).
  Interventions: Behavioral: Stress Management

INTERVENTIONS:
Behavioral: Exposure-Based Treatment for Perfectionism — Three tasks focused on exposures are completed. Each treatment session is approximately twenty minutes.
  Arms: Exposure-Based Treatment for Perfectionism
Behavioral: Stress Management — Videos focused on education about healthy habits and relaxation. Each session is approximately twenty minutes.
  Arms: Stress Management Condition

SUMMARY:
This study is examining the efficacy of a computerized, exposure-based, intervention for perfectionism.

DETAILED DESCRIPTION:
The aim of this study is to further test the efficacy of a short-term, computerized exposure-based treatment for perfectionism (ETP) by comparing it to a stress management condition. ETP consists of three tasks in which participants will repeatedly make mistakes during eight sessions over a two-week period (one session every 2 days).

ELIGIBILITY:
Inclusion Criteria:

- Score of at least 29 on the Frost Multidimensional Perfectionism Scale- Concern over Mistakes subscale

Exclusion Criteria:

* Currently participating in psychotherapy
* Any changes to psychotropic medications in the past four weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse R Cougle, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Department of Psychology, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Clark SA, Patel TA, Cougle JR. Is repeated mistake-making an effective treatment strategy for perfectionism? Findings from a randomized controlled trial. J Behav Ther Exp Psychiatry. 2024 Sep;84:101964. doi: 10.1016/j.jbtep.2024.101964. Epub 2024 May 1. PMID 38704973

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exposure-Based Treatment for Perfectionism | Stress Management Condition
Started | 43 | 42
Completed | 35 | 35
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exposure-Based Treatment for Perfectionism | Stress Management Condition | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.02 (6.65) | 27.69 (7.83) | 27.36 (7.23)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 22 | 17 | 39
  Nonbinary | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black (Not Hispanic) | 7 | 7 | 14
  Race/Ethnicity: White (Not Hispanic) | 22 | 27 | 49
  Race/Ethnicity: Hispanic | 12 | 6 | 18
  Race/Ethnicity: Asian or Pacific Islander | 0 | 1 | 1
  Race/Ethnicity: Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 43 | 42 | 85

OUTCOME MEASURES:

1. Primary Outcome: Frost Multidimensional Perfectionism Scale (FMPS)- Concern Over Mistakes Subscale
Description: Self-report questionnaire examining levels of perfectionism. The concern over mistakes sub-scale includes 9 items with scores ranging from 9 to 45 (higher scores signify higher levels of perfectionism).
Time Frame: Baseline, post treatment (2 weeks), and follow-up (6 weeks)
Population: Number of participants differed at each time point due to drop out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exposure-Based Treatment for Perfectionism | Stress Management Condition
Number analyzed (Participants) | 42 | 42
units on a scale
  Baseline | 34.00 (5.21) | 35.71 (5.25)
  Post-Test: number analyzed (Participants) | 37 | 38
  Post-Test | 34.53 (7.19) | 32.34 (5.97)
  Follow-Up | 32.33 (6.78) | 32.58 (4.96)

2. Secondary Outcome: Center for Epidemiological Studies Depression Scale (CES-D)
Description: Self-report measure used to assess depressive symptoms. Total scores range from 0 to 60 with higher scores indicating a higher level of depressive symptoms.
Time Frame: Baseline, post treatment (2 weeks), and follow-up (6 weeks)
Population: Number of participants differed at each time point due to drop out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exposure-Based Treatment for Perfectionism | Stress Management Condition
Number analyzed (Participants) | 42 | 42
units on a scale
  Baseline | 22.55 (11.20) | 26.45 (11.78)
  Post-Test: number analyzed (Participants) | 37 | 38
  Post-Test | 21.55 (8.61) | 20.63 (10.52)
  Follow-Up: number analyzed (Participants) | 35 | 35
  Follow-Up | 22.17 (11.43) | 20.89 (10.06)

3. Secondary Outcome: Generalized Anxiety Disorder-7
Description: Self-report measure used to assess generalized anxiety symptoms. Scores range from 0 to 21 with higher scores indicating higher levels of generalized anxiety.
Time Frame: Baseline, post treatment (2 weeks), and follow-up (6 weeks)
Population: Number of participants differed at each time point due to drop out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exposure-Based Treatment for Perfectionism | Stress Management Condition
Number analyzed (Participants) | 42 | 42
units on a scale
  Baseline | 9.76 (5.56) | 10.48 (5.12)
  Post-Test: number analyzed (Participants) | 37 | 38
  Post-Test | 9.05 (5.64) | 8.61 (4.78)
  Follow-Up: number analyzed (Participants) | 35 | 35
  Follow-Up | 8.97 (5.41) | 7.56 (4.63)

4. Secondary Outcome: Social Phobia Inventory (SPIN)
Description: Self-report scale that measures social anxiety symptoms. Scores range from 0 to 68 with higher scores indicating higher levels of social anxiety symptoms.
Time Frame: Baseline, post treatment (2 weeks), and follow-up (6 weeks)
Population: Number of participants differed at each time point due to drop out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exposure-Based Treatment for Perfectionism | Stress Management Condition
Number analyzed (Participants) | 42 | 42
units on a scale
  Baseline | 32.79 (15.79) | 34.79 (16.27)
  Post-Test: number analyzed (Participants) | 37 | 38
  Post-Test | 31.12 (19.13) | 28.74 (15.16)
  Follow-Up: number analyzed (Participants) | 35 | 35
  Follow-Up | 30.23 (17.91) | 26.31 (15.19)

5. Secondary Outcome: ED-15
Description: Self-report scale that measures eating disorder symptoms. Scores range from 0 to 6, with higher mean scores indicating higher levels of eating disorder symptoms.
Time Frame: Baseline, post treatment (2 weeks), and follow-up (6 weeks)
Population: Number of participants differed at each time point due to drop out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exposure-Based Treatment for Perfectionism | Stress Management Condition
Number analyzed (Participants) | 42 | 42
units on a scale
  Baseline | 2.84 (1.63) | 2.53 (1.54)
  Post-Test: number analyzed (Participants) | 37 | 38
  Post-Test | 2.41 (1.47) | 2.24 (1.31)
  Follow-Up: number analyzed (Participants) | 35 | 35
  Follow-Up | 2.31 (1.52) | 2.05 (1.31)

6. Secondary Outcome: Irrational Procrastination Scale
Description: Self-report scale that measures levels of procrastination. Scores range from 9 to 45 with higher scores indicating higher levels of procrastination.
Time Frame: Baseline, post treatment (2 weeks), and follow-up (6 weeks)
Population: Number of participants differed at each time point due to drop out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exposure-Based Treatment for Perfectionism | Stress Management Condition
Number analyzed (Participants) | 42 | 42
units on a scale
  Baseline | 25.60 (6.91) | 26.62 (6.97)
  Post-Test: number analyzed (Participants) | 37 | 38
  Post-Test | 23.84 (7.43) | 26.58 (7.18)
  Follow-Up: number analyzed (Participants) | 35 | 35
  Follow-Up | 22.40 (6.07) | 25.11 (6.29)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Exposure-Based Treatment for Perfectionism | Stress Management Condition
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT05351710/Prot_SAP_000.pdf